CLINICAL TRIAL: NCT05095948
Title: Mapping the Processes of Cancer Care Delivery at a Comprehensive Cancer Center
Brief Title: Improving Processes of Cancer Care Delivery at a Comprehensive Cancer Center
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0246; NCI-2021-10266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0246 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-10-12; First posted 2021-10-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Supportive Care (questionnaire, clinic conversation): Patients complete questionnaires over 15-20 minutes and undergo audio recording of clinic conversations between the oncology team or the specialist palliative care team. Patients' medical records are also reviewed.
  Interventions: Procedure: Discussion; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Discussion — Undergo audio recording of clinic conversations
  Other Names: Discuss
Other: Electronic Health Record Review — Review of medical records
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines how cancer care is delivered in oncology and supportive care clinics. Collecting patient feedback may help doctors better understand the processes of cancer care in oncology and supportive care clinics.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the total amount of follow-up clinic time spent on discussing supportive/palliative care issues between primary palliative care provided by the oncology team and specialist palliative care.

SECONDARY OBJECTIVES:

I. To compare between the specialist palliative care team and the oncology team the following aspects of supportive/palliative care delivery: Ia. The number of supportive/palliative care needs the patient reported before the clinic visit (SPARC).

Ib. The number of supportive/palliative care needs the patient wanted to discuss with the clinical team before the clinic visit (SPARC).

Ic. The number of supportive/palliative care needs that were actually raised by the patient during the clinic visit (audiotape).

Id. The number of supportive/palliative care needs that were actually discussed by the clinical team during clinic visit (audiotape).

Ie. The number of supportive/palliative care needs that were documented in progress note by the clinical team after each visit (electronic health record).

If. The number of supportive/palliative care needs that the patient reported had been adequate addressed after the clinic visit (SPARC).

II. To compare the amount of clinic time (both absolute and proportion) spent on discussing supportive/palliative care issues by individual disciplines (e.g. medical doctor, registered nurse, counselor, pharmacist, psychologist, social worker, and priest) between the specialist palliative care team and the oncology team.

III. To examine the nature of topics discussed by the specialist palliative care team and the oncology team and compare the amount of clinic time (both absolute and proportion) spent on each supportive/palliative care issue.

IV. To compare the number of empathic statements between the specialist palliative care team and the oncology team.

V. To compare the processes of supportive/palliative care delivery between patients seeing the oncology team without specialist palliative care (Cohort A) and patients seeing the oncology team when specialist palliative care team is involved (Cohort B).

OUTLINE:

Patients complete questionnaires over 15-20 minutes and undergo audio recording of clinic conversations between the oncology team or the specialist palliative care team. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Within 6 months of diagnosis of metastatic (or stage IV) solid malignancies
* Age 18 or greater
* English speaking
* Follow-up clinic visit (Supportive Care and Medical Oncology Outpatient Clinics at MD Anderson Cancer Center)
* Medical oncologist listed as the attending physician
* COHORT A (Oncology team only cohort): Patients should not have been referred to palliative care services at MD Anderson Cancer Center
* COHORT B (Oncology team and specialist palliative care cohort): Patients should have an upcoming specialist palliative care follow-up visit within 1 week of a medical oncology visit

Exclusion Criteria:

* Delirium (Memorial Delirium Assessment Scale [MDAS] >= 13/30)
* Significant hearing impairment requiring multiple repetitions during the screening process (that may prolong clinic time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients within 6 months of diagnosis of metastatic (or stage IV) solid malignancies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Minutes spent in discussion | through study completion, an average of 1 year
  Will be examined using linear mixed models (LMMs) with physician as the unit of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org